CLINICAL TRIAL: NCT03536390
Title: A Phase 4, Double-blind, Randomized, Parallel Group, Placebo-controlled Study Of The Efficacy And Safety Of Methylphenidate Hydrochloride (Hcl) Extended Release Chewable Tablet (Erct) In 4-5 Year Old Children With Attention Deficit Hyperactivity Disorder (Adhd)
Brief Title: A 6-week Study to Evaluate the Safety and Efficacy of Methylphenidate HCl ERCT in 4-5 Year Old Children With ADHD
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was cancelled prior to the enrollment of any participants.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B7491017
Record Dates: First submitted 2018-05-04; First posted 2018-05-24 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, parallel group study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): one chewable tablet once daily in morning.
  Interventions: Drug: Placebo
- Methylphenidate Hydrochloride Extended Release Chewable Tablet (Experimental): one chewable tablet once daily in morning.
  Interventions: Drug: Methylphenidate Hydrochloride (HCl) Extended Release Chewable Tablet (ERCT)

INTERVENTIONS:
Drug: Methylphenidate Hydrochloride (HCl) Extended Release Chewable Tablet (ERCT) — Methylphenidate Hydrochloride (HCl) Extended Release Chewable Tablet (ERCT)
  Arms: Methylphenidate Hydrochloride Extended Release Chewable Tablet
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This 6-week study is to determine if the study drug, Methylphenidate Hydrochloride (HCl) Extended-Release Chewable Tablets (ERCT), is safe, tolerable and effective when compared to a sugar pill or placebo in children 4 to 5 years of age with ADHD.

DETAILED DESCRIPTION:
Phase 4 Double-blind, Randomized, Parallel Group, Placebo-controlled Study of the Efficacy And Safety of Methylphenidate Hydrochloride (HCl) Extended Release Chewable Tablets (ERCT) In 4-5 Year Old Children With Attention Deficit Hyperactivity Disorder (ADHD)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female child 4-5 years of age at screening.
2. Signed and dated informed consent provided by the subject's parent/legal and assent of the child (as applicable).
3. Meets DSM-5 criteria for ADHD based on the K-SADS-PL.
4. ADHD RS-IV Preschool-Home Version score at Screening and Baseline >/= 90th percentile for gender and age in >/=1 of the following: hyperactive-impulsive subscale, inattentive subscale, or total score.
5. Peabody Picture Vocabulary Test 4 (PPVT-4)Standard Score >/=70.
6. Child Global Assessment Scale (CGAS) score </= 55.
7. Participation in a school type program (day care, preschool, kindergarten, transitional kindergarten, or elementary school) for at least >/=2 half days of the week for at least 3 months and that is anticipated to continue during the study.
8. History of an adequate course of non medication treatment for ADHD based on investigator judgment or, where such treatments are not available, the severity of the subject's ADHD symptoms are such that medication treatment is deemed necessary by the investigator

Exclusion Criteria:

1. Treated with atomoxetine within 30 days prior to the Baseline.
2. Received any investigational products or devices within 30 days prior to the Baseline visit.
3. History of stimulant nonresponse, intolerability or hypersensitivity to any dose of methylphenidate or other stimulant. If a known allergy to D&C red #30, he/she should not be enrolled in the study.
4. An intelligence quotient (IQ) <70.
5. History of acute or chronic medical or psychiatric condition or cardiac or laboratory abnormality.
6. Less than 5th percentile for height or weight at Screening.
7. History of recent clinically significant self-harming behaviors.

Ages: 48 Months to 69 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-09-19 (Estimated); Primary Completion 2021-04-22 (Estimated); Study Completion 2021-04-22 (Estimated)

PRIMARY OUTCOMES:
Attention Deficit Hyperactivity Rating Scale - IV (ADHD RS-IV) Preschool-Home Version | Basline, 6 Weeks
  Change from Baseline to end of double-blind treatment in the total score of the Attention Deficit Hyperactivity Rating Scale - IV (ADHD RS-IV) Preschool-Home Version

SECONDARY OUTCOMES:
Safety-incidence of treatment emergent adverse events | 6 Weeks
  incidence of treatment emergent adverse events
Change from Baseline in Clinical Global Impression - Severity (CGI-S) score | Baseline, Weeks 1 through 6
  The CGI-S is a one-item scale for the clinician to assess their impression of the severity of a subject's current state of illness relative to clinician's past experience with patients who have the same diagnosis. A subject's severity of mental illness is assessed considering a clinician's total clinical experience using a scale from 1 to 7 defined as: 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; or 7=extremely ill.
Change from Baseline in Clinical Global Impression of Improvement (CGI-I) Scale Score | Baseline, Weeks 1 through 6
  The CGI-I is a one-item scale to compare the subject's current condition to the condition at the Baseline (Day -1) visit using a scale from 1 to 7 defined as: 1=very much improved since the initiation of treatment; 2=much improved; 3=minimally improved; 4=no change from baseline (the initiation of treatment); 5=minimally worse; 6= much worse; 7=very much worse since the initiation of treatment.
ADHD RS-IV Preschool-Home Version Total score | Weeks 1 through 5
  The ADHD RS-IV Preschool Version is an 18-item scale corresponding to the 18 items in the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision criteria that is divided into 2 subscales: hyperactivity/impulsivity and inattentiveness. Each item is scored on a 4-point scale ranging from 0 = never/rarely to 3 = very often.
ADHD RS-IV Preschool-Home Version hyperactivity and inattention subscales scores | Weeks 1 through 6
  The ADHD RS-IV Preschool Version is an 18-item scale corresponding to the 18 items in the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision criteria that is divided into 2 subscales: hyperactivity/impulsivity and inattentiveness. Each item is scored on a 4-point scale ranging from 0 = never/rarely to 3 = very often.
ADHD RS-IV Preschool-School Version Total score | Weeks 3 and 6
  The ADHD RS-IV Preschool - School Version will be completed by the subject's teacher.
ADHD RS-IV Preschool-School Version hyperactivity and inattention subscales scores | Weeks 3 and 6
  The ADHD RS-IV Preschool - School Version will be completed by the subject's teacher.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7491017&StudyName=A+Multi-center%2C+Double-blind%2C+Randomized%2C+Placebo-controlled%2C+Parallel+Group+Study+Evaluating+The+Safety+And+Efficacy+Of+Quillivant+Xr+In+The+Treatment+Of+Pre-school+Aged+Children+With+Adhd
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7491017&StudyName=A+Phase+4%2C+Double-blind%2C+Randomized%2C+Parallel+Group%2C+Placebo-controlled+Study+Of+The+Efficacy+And+Safety+Of+Quillichew+Extended+Release+Chewable+Tablets+%28methylphenidate+Hcl+Extended+Release+Chewable+Tablets+%28erct%29%29++In+4-5+Year+Old+Children+With+Attention+Deficit+Hyperactivity+Disorder+%28adhd%29.
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7491017&StudyName=A+Phase+4%2C+Double-blind%2C+Randomized%2C+Parallel+Group%2C+Placebo-controlled+Study+Of+The+Efficacy+And+Safety+Of+Quillichew+%28methylphenidate+Hydrochloride+%28hcl%29%29+Extended+Release+Chewable+Tablets+%28erct%29+In+4-5+Year+Old+Children+With+Attention+Deficit+Hyperactivity+Disorder+%28adhd%29
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7491017&StudyName=A+Phase+4%2C+Double-blind%2C+Randomized%2C+Parallel+Group%2C+Placebo-controlled+Study+Of+The+Efficacy+And+Safety+Of+Methylphenidate+Hydrochloride+%28hcl%29+Extended+Release+Chewable+Tablet+%28erct%29+In+4-5+Year+Old+Children+With+Attention+Deficit+Hyperactivity+Disorder+%28adhd%29